CLINICAL TRIAL: NCT04187599
Title: Post-market Follow Up Study on Paragon CRT® 100 (Paflufocon D) Rigid Gas Permeable Contact Lenses for Corneal Refractive Therapy for Temporary Myopic Refractive Power Reduction
Brief Title: Post-market Follow Up Study on Paragon CRT® 100 (Paflufocon D)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: TigerMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEC-P012019-CRT100
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, open label, 12 month follow up study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Paragon CRT®100 Contact Lens (Experimental): participants will wear the Paragon CRT®100 lens with a follow up for no less than 12 months.
  Interventions: Device: Paragon CRT®100 Contact Lens

INTERVENTIONS:
Device: Paragon CRT®100 Contact Lens — Paragon CRT® 100 Contact Lenses for Corneal Refractive Therapy are indicated for use in the reduction of myopic refractive error in nondiseased eyes.

SUMMARY:
The main objective of this post market clinical study is to evaluate the effectiveness and safety of the Paragon CRT®100 Contact Lens.

DETAILED DESCRIPTION:
This clinical study has two phases: prospective and retrospective.

Prospective Phase - evaluates the post-market long-term effectiveness and safety of the Paragon CRT® 100 Contact Lenses, for temporary myopic refractive power reduction with minimum 12-month period follow-up.

Retrospective phase - evaluates the post-market long-term safety of the Paragon CRT® 100 Contact Lenses, for temporary myopic refractive power reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient contact lens refraction should fit within the available parameters of the study lenses (spherical power within -4.00D and the cylinder power within 1.50D).
2. Is willing to comply with the wear and visit schedule.
3. Is willing to participate and signed the informed consent form.

Exclusion Criteria:

1. Age under 8 years old
2. Any ocular abnormalities, undergone corneal surgery, or history of ocular trauma, active corneal infections (corneal inflammation), corneal curvature less than 40.00D or more than 46.00D
3. Best corrected visual acuity less than 1.0D
4. Pregnant, lactating or near-pregnancy
5. The eye has the following conditions:

   1. Acute and subacute inflammations or infection of the anterior segment of the eye
   2. Any eye disease, injury, or abnormality that affects the cornea, conjunctiva or eyelids, e.g. dacryocystitis, conjunctivitis, blepharitis and other inflammation, glaucoma, etc.
   3. Severe insufficiency of tears (TBUT≤5s).
   4. Allergy to any ingredient, such as mercury or thimerosal, in a solution which is to be used to care
   5. Any active corneal infection (bacterial, fungal or viral).
6. Manifested strabismus
7. Abnormal intra-ocular pressure
8. Suffering from systemic diseases, resulting in low immunity, or affecting corneal re-shaping (such as acute and chronic sinusitis, diabetes, Down syndrome, rheumatoid arthritis, mental patients, etc.)
9. Under medications or long-term medications that lead to dry eye with clinical signs or affects vision and corneal curvature.
10. Examination result indicate any contraindication or not suitable for OrthoK lens wear
11. Participated in pharmaceutical clinical study 3 months before the date of the screening or participated any other medical devices research study within 30 days of the screening
12. Only eye fulfills inclusion criteria
13. History of any ocular operations
14. Unable to follow investigator's instruction
15. Any other condition not suitable for the study per investigator's judgement

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
product effectiveness | 1 month
  Effectiveness=number of eyes with both uncorrected visual acuity and dioptric power meet the "effective" standards/total number of eyes evaluated*100%
uncorrected visual acuity | At baseline
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | 1 day
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 1 week
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 2 weeks
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 1 month
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 3 months
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 6 months
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 9 months
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
uncorrected visual acuity | At 12 months/final visit
  Use standard LogMAR chart to measure the distant uncorrected visual acuity. Use 5.0 system to record LogMAR visual acuity
The dioptric power of subject | At Baseline
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 1 day
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 1 week
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 2 weeks
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 1 month
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 3 months
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 6 months
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 9 months
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The dioptric power of subject | At 12 months/final visit
  Measure dioptric power (subjective dioptric power): include spherical power, cylindrical power, and cylindrical axis
The relevant important parameters of corneal topography of subject | At Baseline
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 1 day
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 1 week
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 2 weeks
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 1 month
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 3 months
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 6 months
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 9 months
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.
The relevant important parameters of corneal topography of subject | At 12 months/final visit
  The corneal topographer is used for measurement, and the relevant parameters include: corneal curvature on the steep meridian Ks, corneal curvature on the flat meridian Kf, and corneal astigmatism.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Jun, MD, Principal Investigator — The Affiliated Eye Hospital of Wenzhou Medical University; Qu Xiao Mei, MD, Principal Investigator — Eye & ENT Hospital of Fudan University; Yang Zhi Kuan, MD, Principal Investigator — Changsha Aier Eye Hospital; Li Li Hua, MD, Principal Investigator — Tianjin Eye Hospital
Locations (4):
- China (4):
  - Changsha Aier Eye Hospital, Shanghai
  - Eye & ENT Hospital of Fudan University, Shanghai
  - Tianjin Eye Hospital, Tianjin
  - The Affiliated Eye Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No